CLINICAL TRIAL: NCT06456151
Title: Invasive Candidiasis in Critical Care
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: University Hospital, Motol (Other)
Responsible Party: Sponsor
Other Study IDs: ULM-01-Invasive candidiasis; 03/RVO-FNOs/2024 (Other Grant/Funding Number: University Hospital Ostrava); SGS06/LF/2024 (Other Grant/Funding Number: Faculty of Medicine, University of Ostrava)
Record Dates: First submitted 2024-06-04; First posted 2024-06-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Invasive Candidiasis
Keywords: invasive candidiasis; biomarkers; candida sepsis
MeSH Terms: conditions — Candidiasis, Invasive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Left-over blood samples from patients will be used in the study. The study subjects will be also asked for a sample of urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected invasive candidiasis: Patients with suspected invasive candidiasis will be enrolled in this study arm.
  Interventions: Diagnostic Test: Invasive candidiasis test; Other: Urine sample collection for future research

INTERVENTIONS:
Diagnostic Test: Invasive candidiasis test — The combination of acute phase marker monitoring and the T2Candida assay will be assessed.
Other: Urine sample collection for future research — Patients will be asked to provide a urine sample for future research (urine biobank).

SUMMARY:
The combination of acute phase marker monitoring and the "T2Candida" assay (name of the test) will represent an acceleration of the identification of the causative agent of mycotic infection, a significant improvement in the specificity and positive predictive value of this strategy in the diagnosis of invasive candidiasis and candidemia in ICU patients, thereby improving the clinical condition of patients and reducing the cost of specific antifungal therapy.

DETAILED DESCRIPTION:
Speed of response in the treatment of sepsis is crucial for the patient. The time from the collection of a positive haemoculture to the identification of the causative agent of sepsis is around 2 days; therefore, physicians in intensive care units deploy combined empiric antibiotic and antifungal therapy immediately when acute phase markers such as procalcitonin, interleukin-6, Presepsin, C-reactive protein are elevated. A new acute phase marker is lipopolysaccharide-binding protein, which, together with Presepsin, appears to be a suitable marker to distinguish invasive candida infections from bacterial infections. But its kinetics needs to be further analyzed.

At the same time, the causative agent of sepsis, G-/G+ bacteria or yeast, must be identified as soon as possible. Haemoculture and culture of the established drain is the gold standard, but the disadvantage is the low sensitivity and the time delay to obtain the result. It is therefore advisable to combine haemoculture with molecular biology-based tests that can identify the causative organism within hours. Conversely, the disadvantage of these tests is that they identify only the most common sepsis pathogens and do not determine susceptibility to antibiotics and antifungals, but the advantage is that with prophylaxis in place, these tests are often positive when haemoculture is negative. The T2Candida test can detect Candida albicans, Candida tropicalis, Candida glabrata, Candida krusei and Candida parapsilosis, which are the more common causative agents of mycotic bloodstream infections.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients
* new onset sepsis
* rise in body temperature >38°C according to The Third Consensus Definitions for Sepsis and Septic Shock
* colonization with Candida spp. from more than 1 non-sterile site
* body temperature >38 °C despite 5 days of broad-spectrum antibiotic therapy with the presence of at least 1 of the following risk factors: abdominal surgery, secondary peritonitis, pancreatitis, central venous catheter (CVC) insertion, total parenteral nutrition (CPV), dialysis, steroid therapy, immunosuppressive therapy, or liver transplantation
* microbiological test results will be reviewed and categorized based on whether Candida sp. is isolated from at least 2 non-sterile sites (±3 days) and whether there is an alternative microbiological diagnosis.

Exclusion Criteria:

* not signing the informed consent with participation in the study
* administration of antifungal therapy prior to collection of the biological material required for the study

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected invasive candidasis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Acute-phase biomarkers dynamics - procalcitonin | 8 days
  The levels of procalcitonin will be observed in time and measured in μg/L. The follow-up will last 8 days, the patient may be observed repeatedly, depend-ing on the patient's condition.
Acute-phase biomarkers dynamics - interleukin-6 | 8 days
  The levels of interleukin-6 will be observed in time and measured in pg/ml. The follow-up will last 8 days, the patient may be observed repeatedly, depend-ing on the patient's condition.
Acute-phase biomarkers dynamics - interleukin-10 | 8 days
  The levels of interleukin-10 will be observed in time and measured in pg/ml. The follow-up will last 8 days, the patient may be observed repeatedly, depend-ing on the patient's condition.
Acute-phase biomarkers dynamics - Presepsin | 8 days
  The levels of Presepsin will be observed in time and measured in pg/ml. The follow-up will last 8 days, the patient may be observed repeatedly, depend-ing on the patient's condition.
Acute-phase biomarkers dynamics - C-reactive protein | 8 days
  The levels of C-reactive protein will be observed in time and measured in mg/dL.
  The follow-up will last 8 days, the patient may be observed repeatedly, depend-ing on the patient's condition.
Acute-phase biomarkers dynamics - 1,3-β-D-glucan | 8 days
  The levels of C-reactive protein will be observed in time and measured in pg/ml.
  The follow-up will last 8 days, the patient may be observed repeatedly, depend-ing on the patient's condition.
Acute-phase biomarkers dynamics - pentraxin 3 | 8 days
  The levels of C-reactive protein will be observed in time and measured in ng/ml.
  The follow-up will last 8 days, the patient may be observed repeatedly, depend-ing on the patient's condition.
T2Candida test | One-time measurement at the enrolment into the study
  The T2Candida test is able to detect the presence of Candida albicans, C. tropicalis, C. glabrata, C. krusei and C. parapsilosis. The results will be assessed as positive or negative.
Lipopolysaccharide binding protein | One-time measurement at the enrolment into the study
  The levels of Lipopolysaccharide binding protein (LBP)_S/P will be observed in time and measured in mg/L.
  The follow-up will last 8 days, the patient may be observed repeatedly, depend-ing on the patient's condition.

CONTACTS AND LOCATIONS:
Overall Officials: Hana Slepčanová, Mgr., Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Motol, Prague

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Dobias R, Kanova M, Petejova N, Pisti SK, Bocek R, Krejci E, Struzkova H, Cachova M, Tomaskova H, Hamal P, Havlicek V, Raska M. Combined Use of Presepsin and (1,3)-beta-D-glucan as Biomarkers for Diagnosing Candida Sepsis and Monitoring the Effectiveness of Treatment in Critically Ill Patients. J Fungi (Basel). 2022 Mar 17;8(3):308. doi: 10.3390/jof8030308. PMID 35330311
- [Background] Bassetti M, Giacobbe DR, Vena A, Wolff M. Diagnosis and Treatment of Candidemia in the Intensive Care Unit. Semin Respir Crit Care Med. 2019 Aug;40(4):524-539. doi: 10.1055/s-0039-1693704. Epub 2019 Oct 4. PMID 31585478
- See also: World Health Organisation (WHO) fungal priority pathogens list to guide research, development and public health action — https://www.who.int/publications/i/item/9789240060241